CLINICAL TRIAL: NCT04213508
Title: Isotonic vs Hypertonic Nasal Irrigation and Frequency of Irrigation Per Day in Rhinosinusitis Patients
Brief Title: Type and Frequency of Nasal Irrigation in Rhinosinusitis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-2019-01-262
Record Dates: First submitted 2019-12-07; First posted 2019-12-30 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Otorhinolaryngologic Diseases; Rhinosinusitis
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Rhinosinusitis | interventions — Sodium Chloride; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind Study ( Both Participants and Investigator are masked ).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Isotonic saline with frequency of 2 times per day (Active Comparator): 0.9% Sodium Chloride (NaCl) saline will be used as nasal irrigation for 2 times per day. Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time) . So, in total 200 ml of 0.9% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Interventions: Drug: Isotonic Saline ( 0.9% Sodium Chloride Saline)
- Hypertonic saline with frequency of 2 times per day (Active Comparator): 3% Sodium Chloride (NaCl) saline will be used as nasal irrigation for 2 times per day. Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time) . So, in total 200 ml of 3% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Interventions: Drug: Hypertonic Saline ( 3% Sodium Chloride Saline)
- Isotonic saline with frequency of 5 times per day (Active Comparator): 0.9% Sodium Chloride (NaCl) saline will be used as nasal irrigation for 5 times per day. Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time) . So, in total 500 ml of 0.9% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Interventions: Drug: Isotonic Saline ( 0.9% Sodium Chloride Saline)
- Hypertonic saline with frequency of 5 times per day (Active Comparator): 3% Sodium Chloride (NaCl) saline will be used as nasal irrigation for 5 times per day. Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time) . So, in total 500 ml of 3% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Interventions: Drug: Hypertonic Saline ( 3% Sodium Chloride Saline)

INTERVENTIONS:
Drug: Isotonic Saline ( 0.9% Sodium Chloride Saline) — 0.9% Sodium Chloride (NaCl) saline will be used as nasal irrigation for two groups. (first groups 2 times per day and second group 5 times per day ). Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time) . So, in total 500 ml of 0.9% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Arms: Isotonic saline with frequency of 2 times per day; Isotonic saline with frequency of 5 times per day
Drug: Hypertonic Saline ( 3% Sodium Chloride Saline) — 3% Sodium Chloride (NaCl) saline will be used as nasal irrigation for two groups. (first groups 2 times per day and second group 5 times per day ). Each time, amount of 50 ml of saline will be used in each nostril ( 100 ml for both nostrils per time). So, in total 200 ml of 3% Sodium Chloride (NaCl) saline will be used daily for 1 month .
  Arms: Hypertonic saline with frequency of 2 times per day; Hypertonic saline with frequency of 5 times per day

SUMMARY:
Rhinosinusitis is a common clinical problem with significant morbidity which alters patients' quality of life that has its effect on 1 out of 7 adults. It has been found that rhinosinusitis accounts for almost 26 million clinics and emergency visits per year in United states .Nasal irrigation is standard management used to treat a variety of sinonasal diseases. Furthermore, nasal irrigation decreases the need of usage other medications in rhinosinusitis .Hence, it is considered safe, inexpensive, and easy to use with no evidence of major adverse effects .Up to our knowledge, there is no clear guideline in which type (isotonic saline vs hypertonic saline) and frequency (times per day) of nasal irrigation are superior and better.

DETAILED DESCRIPTION:
Nasal irrigation is one of the main treatment of sinonasal diseases. The mechanism of action of nasal irrigation has many physiological aspects such as removing of excess mucus which is a potential medium for bacterial growth and infection, cleaning of antigens and biofilm to decrease inflammatory process, increase mucocilliary function and removing curst and debris from post-surgery to enhance wound healing and mucosalization Hypertonic saline is defined as a solution with more than 0.9% weight per volume of sodium chloride while isotonic saline is defined as a solution that equals to 0.9% weight per volume of sodium chloride. There are controversial studies in the literature on which saline is superior on the other, some prefer hypertonic saline over isotonic saline because it can move water outside the cells, decrease edema of mucosa, increase hydration of sol layer and decrease muco-adhesiveness and improve mucociliary clearance while others found both solution had same efficacy, improved nasal stuffiness and nasal obstruction but patients prefer isotonic saline because it is well tolerated and less burning sensation. Frequency of nasal irrigation per day is poorly studied in the literature with no known recommended times per day. Our aim is to find which type of saline and number of irrigation per day are better and statistically significant .

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years of either gender
* Acute and chronic rhinosinusitis

Exclusion Criteria:

* History of nasal or sinus surgery
* Age less than 18 years of either gender
* diagnosis other than rhinosinusitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test 22 . | Change from baseline of Sino-Nasal Outcome Test 22 (SNOT-22) at 1 month
  The Sino-Nasal Outcome Test (SNOT-22) is a validated chronic rhinosinusitis -specific outcome measure consisting of 22 items that captures sinus-specific and general health-related impact of the disease process.
  To answer the instrument, patients suggest their level of affection in each domain and identify the most 5 important items. Each item quantifies symptoms severity from 0 (no problem) to 5 (worst symptom). The sum of each item results in a maximum score of 110 while the minimum is 0 . High score indicates poor outcome.
  Arabic version of a validated and reliable SNOT-22 will utilize in this study. We will measure the change of SNOT-22 from our baseline after follow up in 1 month
Change in Peri-Operative Sinus Endoscopy Score | Change from baseline of Peri-Operative Sinus Endoscopy (POSE) at 1 month
  Peri-Operative Sinus Endoscopy Score (POSE) is objective endoscopic scoring system was utilized to assess the surgical outcomes in the sinonasal cavities through the evaluation of the middle turbinate, middle meatal antrostomy,ethmoid cavity, and secondary sinuses.The sum of maxiumum score is 20 while the minimum is 0 . High score indicates poor result . Th We will measure the change of POSE from our baseline after follow up in 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad H Albar, MD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- Imam abdulrahman bin faisal university, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided